CLINICAL TRIAL: NCT06700421
Title: A Prospective, Single-center, Phase II Clinical Study of Adebrelimab Combined with Apatinib in the Treatment of Unresectable Stage III NSCLC Patients with Grade ≤2 Radiation Pneumonitis After Definitive Chemoradiotherapy
Brief Title: Phase II Clinical Study of Adebrelimab Combined with Apatinib in the Treatment of Locally Advanced Non-small Cell Lung Cancer Patients with Radiation Pneumonitis
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Wei Zhou (Other)
Responsible Party: Sponsor-Investigator, Wei Zhou, Director of Radiation Oncology Center, Chongqing University Cancer Hospital
Organization: Chongqing University Cancer Hospital (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MA-NSCLC-II-035
Record Dates: First submitted 2024-11-20; First posted 2024-11-22 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-11

CONDITIONS: Unresectable Locally Advanced Non-small Cell Lung Cancer
Keywords: Unresectable locally advanced non-small cell lung cancer; Radiation pneumonitis; Adebrelimab; Apatinib; Chemoradiotherapy
MeSH Terms: conditions — Radiation Pneumonitis | interventions — apatinib; Immunotherapy; Immune Checkpoint Inhibitors; Angiogenesis Inhibitors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A (Other): Patients with grade 0-1 radiation pneumonitis were enrolled and treated with adebrelimab combined with apatinib within 42 days after definitive chemoradiotherapy
  Interventions: Drug: Adebrelimab + Apatinib
- Group B (Other): Patients with grade 2 radiation pneumonitis were enrolled and treated with adebrelimab combined with apatinib within 56 days after definitive chemoradiotherapy
  Interventions: Drug: Adebrelimab + Apatinib

INTERVENTIONS:
Drug: Adebrelimab + Apatinib — Adebrelimab combined with apatinib
  Other Names: immunotherapy; Programmed death ligand 1 inhibitor; Antiangiogenic agents

SUMMARY:
A prospective, single-center, phase II clinical study of adebrelimab combined with apatinib in the treatment of unresectable stage III NSCLC patients with grade ≤2 radiation pneumonitis after definitive chemoradiotherapy

DETAILED DESCRIPTION:
A prospective, single-center, phase II clinical study of adebrelimab combined with apatinib in the treatment of unresectable stage III NSCLC patients with grade ≤2 radiation pneumonitis after definitive chemoradiotherapy.At least 32 participants will be enrolled in this study.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years old, male or female;
2. ECOG PS score 0-1;
3. The expected survival time is not less than 12 weeks;
4. Histologically or cytologically confirmed non-small cell lung cancer patients with unresectable locally advanced (stage III) (AJCC TNM staging, 8th edition);
5. Patients who are not candidates for EGFR, ALK, or ROS1 targeted therapy, as confirmed by histologic or cytologic specimens (with documented evidence of no EGFR sensitizing mutation, ALK gene rearrangement, or ROS1 gene fusion);
6. Patients with grade 2 or below radiation pneumonitis without disease progression after receiving platinum-based concurrent/sequential chemoradiotherapy;
7. First dose was administered on days 1-42 (up to 42 days) after completion of concurrent/sequential platinum-based chemoradiotherapy for grade ≤1 RP; Patients with grade 2 RP who were downgraded to less than grade 1 RP within 56 days (including 56 days) after concurrent/sequential chemoradiotherapy received the first medication, and consolidation chemotherapy after radiotherapy was not allowed during the period.

All toxic effects from previous antineoplastic therapy, except hearing loss, alopecia, and fatigue, had to have recovered to grade 1 or less (according to NCI CTCAE V5.0) or baseline levels to be eligible.

9. Have not received any anti-CTLA-4, anti-PD-1, anti-PD-L1/2, anti-angiogenesis inhibitors, or anti-tumor vaccine therapy; 10. Provide or collect biopsy tissue or blood samples during the treatment for biomarker analysis according to the subjects' wishes; 11. Normal function of major organs and bone marrow; 12. Female subjects of childbearing potential had to have a negative serum or urine pregnancy test 72 hours before starting the trial and be willing to use a highly effective, medically approved contraceptive method for the duration of the study and for 90 days after the last dose of the trial drug; Male participants whose partner was a woman of childbearing potential agreed to use an effective method of contraception or to be surgically sterilized for the duration of the study and for 90 days after the last dose of the trial drug.

13. The subjects voluntarily participated in this study, and signed the informed consent form. The compliance was good, and the efficacy and adverse reactions were followed up according to the protocol.

Exclusion Criteria:

1. Histological types of mixed small cell lung cancer and non-small cell lung cancer;
2. Disease progression after chemoradiotherapy; Had undergone major surgery within 28 days before the first dose of a study drug or was planned to undergo major surgery during the study (at the investigator's discretion); 3.

4. Administration of live attenuated vaccine within 28 days prior to dose or planned for the duration of the study; 5. Participated in another clinical study within 28 days before the first use of a trial drug, and used any trial drug; 6. Grade ≥3 radiation pneumonitis caused by chemoradiotherapy; 7. Imaging (CT/MRI) showed that the tumor invaded the large blood vessels or had unclear boundaries with blood vessels; 8. Known history of allogeneic organ transplantation or allogeneic hematopoietic stem cell transplantation; 9. Presence of any active autoimmune disease or a history of autoimmune disease with expected recurrence; 10. Congenital or acquired immune deficiency; 11. Suffering from an infectious disease that is poorly controlled; 12. Subjects requiring systemic treatment with corticosteroids (>10mg/ day of prednisone or equivalent dose of the same hormone) or other immunosuppressive agents within 14 days before the first dose of the trial drug; 13. Cancer other than NSCLC in the past 5 years; 14. Evidence of past or current severe impairment of lung function, with forced expiratory volume in 1 second (FEV1) <1.2L or DLCO<50% of predicted value; 15. Grade II or above myocardial ischemia or myocardial infarction with poorly controlled arrhythmia; 16. Have poorly controlled hypertension; 17. Occurrence of arterial/venous thrombotic events (cerebral embolism, deep vein thrombosis, pulmonary embolism, etc.) within 6 months before the first dose; 18. Subjects with clinically significant bleeding symptoms or clear evidence or history of bleeding tendency within 3 months before the first dose; 19. Obvious hemoptysis symptoms within 30 days before the first dose or hemoptysis of 2.5mL or more per day; 20. Known hereditary or acquired bleeding and thrombophilia (e.g. hemophilia, coagulopathy, thrombocytopenia, hypersplenism, etc.); 21. Urine routine showed urine protein ≥ (++), or 24-hour urine protein ≥ 1.0g; 22. The need for systemic antibiotics due to infection within 14 days before the first dose of medication; Or unexplained fever > 38.5 ° C 14 days before the first dose of medication; 23. Pregnant or lactating women; 24. Known allergy or intolerance to the study drug or its excipients; 25. Any condition that the investigator considers may harm the subject or cause the subject to be unable to meet or perform the requirements of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2024-08-13 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression free survival (PFS) | Doses were administered every 6 weeks from the first dose of study drug until approximately 12 months
  Refers to the time from the start of nonrandomization until tumor progression or death from any cause, whichever occurs first

SECONDARY OUTCOMES:
overall survival, OS | Doses were administered every 6 weeks from the first dose of study drug until approximately 12 months
  Refers to the time from the start of nonrandomization until death from any cause.
Objective Response Rate, ORR | Doses were administered every 6 weeks from the first dose of study drug until approximately 12 months
  Refers to the proportion of patients who have achieved a pre-defined tumor volume reduction (CR/PR) and maintained the minimum time frame required by the accepted response evaluation criteria (such as solid tumor RECIST Version 1.1).
Disease control rate, DCR | Doses were administered every 6 weeks from the first dose of study drug until approximately 12 months
  Proportion of all subjects whose best overall response (BOR) was rated as complete response (CR), partial response (PR), and stable disease (SD) according to RECIST v1.1 criteria.
Duration of response, DOR | Doses were administered every 6 weeks from the first dose of study drug until approximately 12 months
  Defined as the period from the date the tumor remission was first recorded to the date the disease progression was first recorded or the date of death from any cause

CONTACTS AND LOCATIONS:
Overall Officials: Wei Zhou, Principal Investigator — Chongqing University Cancer Hospital
Locations (1):
- Chongqing University Cancer Hospital, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
The survival data of individual participant will be shared after the research iscompleted.
Supporting Information: Study Protocol, CSR
Time Frame: After the study is completed.
Access Criteria: Other Medical Professionals with permission from Principle Investigator